CLINICAL TRIAL: NCT01150318
Title: Study of the Testicular Function After Iodine 131 Therapy in Patients With Papillary Carcinoma
Brief Title: Testicular Function After Iodine 131 Therapy in Papillary Carcinoma Patients
Acronym: SAPIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe Aucan, Department Clinical Research of Developpement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P040419
Record Dates: First submitted 2010-04-29; First posted 2010-06-24 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Thyroid Neoplasms
Keywords: Male; Infertility; Radioisotopes Therapy; Follicular thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Infertility; Adenocarcinoma, Follicular | interventions — Iodine-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients treated by 131 iodine for thyroid cancer
  Interventions: Drug: Administration of 131 iodine

INTERVENTIONS:
Drug: Administration of 131 iodine — 100 mCi 131 iodine irradiation
  Other Names: 131 iodine

SUMMARY:
Papillary cancer may affect patients of any age,with a good prognosis. Most of young patients may hence procreate as often as the general population.131iodine is an essential tool during treatment of thyroid cancer. According literature data, 131iodine given patients may experience exocrine testicular dysfunction with transient azoospermia, as a significant growing number of Desoxyribonucleic acid (DNA) damage may concern the patient or his offspring. The primary purpose will be to study a genomic instability within the germinal line, based on a significant mutation rate analysis in their minisatellites regions after 100 mCi 131 iodine irradiation compared to the baseline spermogram of each patient, thus being his own control case in a cross-over study.The inclusion of 50 patients treated by surgery prior to131iodine would result in statistically significant results.This multicentric cross-over study with a multidisciplinary approach will act for a direct benefit on testis function in patients aged 18-45 treated by 131iodine for thyroid cancer. Samples measurements timing will be: after surgery, 2 and 12 months after 131iodine administration.

DETAILED DESCRIPTION:
Papillary cancer may affect patients of any age,with a good prognosis. Most of young patients may hence procreate as often as the general population.

131iodine is an essential tool during treatment of thyroid cancer, concerning ablation of the orthotopic thyroid remnant and/or distant metastasis. According literature data, 131iodine given patients may experience exocrine testicular dysfunction with transient azoospermia, as a significant growing number of DNA damage may concern the patient or his offspring. No higher malformation risk has been described in children fathered by patients who has received 131iodine for thyroid cancer. But animal studies showed a genomic instability leading to a major cancer risk in the offspring of male mice receiving isotopic radiotherapy. The deduced hypothesis is that a genetic toxicity of those radiation exists on the germ cells, and most of all that those acquired mutations may be transmitted to the next generation, majoring a risk of somatic mutation accumulation. So is described TCHERNOBYL exposed patients and their children. Unfortunately, little is known on trans-generational genomic instability.

The primary outcome will be to study a genomic instability within the germinal line, based on a significant mutation rate analysis in their minisatellite regions after 100 mCi 131 iodine irradiation compared to the baseline spermogram of each patient, thus being his own control case in a cross-over study. Literature reports a risk ratio rising from 1,4 to 1,6 for a comparable exposition dose. Under a 2,5 % spontaneous mutation rate hypothesis and for 1000 minisatellites studied per subject, with the mutation rate rising to 50% (RR=1,5), as the inter-individual variability is expected to be high : the inclusion of 50 patients treated by surgery prior to131iodine would result in statistically significant results.

Secondary outcomes will be to look for deleterious endpoints on spermatogenesis, such as : apparition of a low number of spermatozoids, a low vitality, a low mobility, elevated apoptosis and aneuploidy rate found in sperm of treated subjects vs before iodine treatment. Therefore, the kinetics of spermogram parameters alteration will be available. Testosterone/LH ratio will be assessed before and after 131iodine. Direct measure of testis irradiation obtained by a scrotal dosimeter will permit calculation of the delivered irradiation dose and a dose/effect relation between the different parameters.

This multicentric cross-over study with a multidisciplinary approach will act for a direct benefit on testis function in patients aged 18-45 treated by 131iodine for thyroid cancer. Samples measurements timing will be: after surgery, 2 and 12 months after 131iodine administration. Therefore, endpoints such as medical examination, exocrine and endocrine testis function in blood and spem sampling will be assessed in order to obtain spermogram, Sperm Cytogram, aneuploidy/apoptosis, minisatellites region mutation rate. Medical examination will take place in each local site, either from endocrinology, oncology, nuclear medicine departments. The sperm samples and spermogram, Sperm Cytogram, irradiation- induced abnormalises studies will be centralized at the CECOS (Tenon Hospital, Paris, France). Hormonal dosages will be processed in Bicetre Hospital (Kremlin-Bicetre, France). Minisatellites mutations study processed on frozen sperm samples will take place in the Genetic of Radiosensibility Department (Commissionership in the energy atomic, SACLAY, France).

This study would permit to measure out the minisatellites region mutation rate frequency, aneuploidy and DNA damage frequency, and finally kinetics of those alterations after 131iodine irradiation for human thyroid cancer. At the clinical level, practitioners would more precisely advise their patients on potential fertility risks and help to choose the appropriate practice in order to preserve it before thyroid cancer treatment. Knowing those results, it may redefine iodine indication. The knowledge of irradiation-induced genomic abnormalises is critical, regarding the growing number of examinations (Computed Tomography or Positron Emission Tomography-scans), known to deliver the same amount of irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Men from 18 to 55 years treated by thyroid surgery for papillary carcinoma followed by iodine 131 radiotherapy
* informed consent

Exclusion Criteria:

* The patients under supervision (guardianship), under guardianship.
* Patients of less than 18 years old and furthermore of 55 years old
* Hypogonadism known or bare during the hormonal balance sheet of inclusion.
* The patients with a history of definitive azoospermia·
* Azoospermia at baseline spermogram
* Chemotherapy or radiotherapy history
* The patients exposed to toxic substance for the spermatogenesis

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
A genomic instability within the germinal line | 12 months after iodine131 administration
  To study a genomic instability within the germinal line, based on a significant mutation rate analysis in their minisatellite regions after 100 mCi 131 iodine irradiation compared to the baseline spermogram of each patient, thus being his own control case in a cross-over study

SECONDARY OUTCOMES:
The spermatozoid apoptosis and aneuploidy levels | 1 month before iodine131 administration
The exocrine and endocrine testicular function | 1 month before iodine131 administration
The radiation doses delivered to the testis in exposed patients | 72 hours after 131 iodine administration
The exocrine and endocrine testicular function | 3 months after iodine131 administration
The exocrine and endocrine testicular function | 12 months after iodine131 administration
The spermatozoid apoptosis and aneuploidy levels | 3 months after iodine131 administration
The spermatozoid apoptosis and aneuploidy levels | 12 months after iodine131 administration

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bouchard, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Saint Antoine Hospital, Endocrinology Unit, Paris, France

REFERENCES:
- [Derived] Bourcigaux N, Rubino C, Berthaud I, Toubert ME, Donadille B, Leenhardt L, Petrot-Keller I, Brailly-Tabard S, Fromigue J, de Vathaire F, Simon T, Siffroi JP, Schlumberger M, Bouchard P, Christin-Maitre S. Impact on testicular function of a single ablative activity of 3.7 GBq radioactive iodine for differentiated thyroid carcinoma. Hum Reprod. 2018 Aug 1;33(8):1408-1416. doi: 10.1093/humrep/dey222. PMID 29912343